CLINICAL TRIAL: NCT03102099
Title: Application Value of Contrast-enhanced Ultrasound-guided Fine-needle Aspiration Biopsy in the Evaluation of Thyroid Nodules
Brief Title: Contrast-enhanced Ultrasound-guided Fine-needle Aspiration Biopsy in the Evaluation of Thyroid Nodules
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Ying Fu, Principal Investigator, Peking University Third Hospital
Other Study IDs: PekingUTH_001
Record Dates: First submitted 2017-03-10; First posted 2017-04-05 (Actual); Last update posted 2017-04-05 (Actual); Status verified 2017-03

CONDITIONS: Thyroid Nodules
MeSH Terms: conditions — Thyroid Nodule

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- contrast-enhanced ultrasound group: The contrast-enhanced ultrasound(CEUS)patients will undergo biopsy with contrast-enhanced ultrasound guidance.
  Interventions: Procedure: contrast-enhanced ultrasound group
- conventional ultrasound group: The conventional ultrasound group will undergo biopsy with conventional ultrasound guidance.
  Interventions: Procedure: conventional ultrasound group

INTERVENTIONS:
Procedure: contrast-enhanced ultrasound group — The contrast-enhanced ultrasound patients will undergo biopsy with contrast-enhanced ultrasound guidance.
  Groups: contrast-enhanced ultrasound group
Procedure: conventional ultrasound group — The conventional ultrasound group will undergo biopsy with conventional ultrasound guidance.
  Groups: conventional ultrasound group

SUMMARY:
To evaluate the application value of contrast-enhanced ultrasound in the diagnosis of thyroid nodules using fine needle aspiration.

DETAILED DESCRIPTION:
Thyroid nodules and thyroid cancer are common and frequently occurring diseases in China; Relevant researches reveal that the increase in the incidence of thyroid cancer is more prominent in China than that of overseas, the incidence of thyroid cancer in urban residents of Beijing increased from 1.55/100,000 in 1995 to 9.9/100,000 in 2010 (5.38 fold).

The rapid development of imaging techniques including ultrasound, CT and MRI had substantially increased the accuracy in the diagnosis of thyroid nodules, however the accuracy is still not up to 100% and a further aspiration biopsy is required. Therefore, ultrasound-guided percutaneous biopsy plays a critical role in the diagnosis of pathological lesions. Many guidelines deem fine needle aspiration (FNA) biopsy to be the most accurate and cost-effective examination method in the evaluation of thyroid nodules as it helps to reduce unnecessary thyroid nodule surgeries and it also helps the clinicians to determine the appropriate surgical treatment plan[1-4]. However according to literature reports, samples with insufficient quantity of cells can occur up to 10-15% of the cases, sometimes a second biopsy or a diagnostic operation needs to be performed[1,4].False negative results of FNA biopsy or a mismatch between ultrasound diagnosis and clinical diagnosis can occur due to a number of reasons such as the tumor being too big or too small, a poor location, presence of degenerative necrosis, inappropriate position of biopsy or be affected by the operator's experience etc.

Contrast-enhanced ultrasound (CEUS) is a new technology which is recently introduced into China, it has the ability to display the microvascular perfusion of the tissue under a low mechanical index. The serial real-time images obtained can be digitalized and dynamically stored. And this allows for retrospective analysis and also enables comparison to be made with other imaging techniques. CEUS can sensitively reflect the characteristics of blood supply and microcirculation at the site of the lesion.

Although CEUS-guided FNA of thyroid nodules has not yet been reported, a large number of studies have reported liver biopsy performed under the guidance of CEUS. Its efficacy in obtaining accurate diagnosis and in reducing the number of biopsies is clear when samples are taken from the area of rich blood supply.

Metabolic-active areas within the malignant tumor, or areas of degeneration or necrosis and also the detection of small tumors can be confirmed through the use of CEUS. Aspiration biopsy when performed under the guidance of CEUS is expected to yield decreased non-diagnostic result. The investigators intent to create a randomized controlled study to investigate the application value of CEUS in the diagnosis of space-occupying lesions of the thyroid using FNA.

Data collection Collect and sort out the general data of patients, record the conventional US findings and the contrast-enhanced ultrasound (group CEUS) findings of the two groups, and also the results from aspiration biopsy and pathology, fill in the case report form (CRF), establish a database. Carry out analysis using specialized statistical software. Four parameters of efficacy (inadequacy, indeterminacy, malignancy, and benign) rates) were evaluated in the series of thyroid FNA and compared with the two groups. The inadequacy rate refers to the proportion of cases with a non-diagnostic result. The indeterminate rate refers to the proportion of cases with an atypia of undetermined significance/follicular lesion of undetermined significance (AUS or FLUS) category. The malignancy rate refers to the proportion of cases that were malignant. The benign rate refers to the proportion of cases that were benign. The number of obtained cells in the specimens with diagnostic result was classified into two classes according the cytopathologist's experience: intermediate (diagnosed possible), and abundant (diagnosed easily). The comparison of cell amount between the two groups is secondary aim.

Statistical analysis Statistical analysis is carried out using SPSS 22.0, all statistical data will be analyzed using the Chi square test. Differences were considered statistically significant at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a space-occupying thyroid lesion found either via conventional ultrasound or CT/MRI and clinically requiring a further biopsy.
* Age 18 years old or above with no limitation of gender.
* Obtain a signed informed consent.

Exclusion Criteria:

* Contraindications to the use of contrast agents as described by the medication guide.
* Patients who are contraindicated to aspiration biopsy: patients with unexplained bleeding history, severe anemia, or patients who have a tendency to bleed and this bleeding disorder has not been corrected (prothrombin time 3-5seconds longer than the normal control, platelet count <60000/mm3); no safe aspiration path; menstruating female patients.
* If the patient has a serious psychological or mental problem, and is suspected to have a poor compliance with the current clinical study, or maybe unable to obtain a definitive diagnosis for the lesion.
* Pregnant or lactating women or women with a positive pregnancy test before their first medications are given.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who intends to perform fine needle aspiration (FNA) at the Peking University Third hospital.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2018-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
The Bethesda System for Reporting Thyroid Cytology (TBSRTC) | From date of randomization until the date of first documented cytopathology result of fine needle aspiration (FNA) on the suspected nodule, assessed up to 1 month
  To evaluate contrast-enhanced ultrasound (CEUS) improving the technical sufficiency of fine needle aspiration (FNA). The Bethesda System for Reporting Thyroid Cytology (TBSRTC) has six general diagnostic categories. Each of the categories has an implied cancer risk (ranging from 0 to 3% for the benign category to nearly 100% for the malignant category) with rational clinical management guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Fu, Ph.D, Principal Investigator — Peking University Third Hospital; Li-Gang Cui, M.D., Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided